CLINICAL TRIAL: NCT00134329
Title: Erectile Dysfunction and Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Other Study IDs: 2005/096
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus; Erectile Dysfunction
MeSH Terms: conditions — Diabetes Mellitus; Erectile Dysfunction

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Filling out a questionnaire on the possible occurrence of erectile dysfunction

SUMMARY:
This study consists of filling out a questionnaire on possible erectile dysfunction.

DETAILED DESCRIPTION:
Male diabetic patients who attend a diabetic routine year program visit will be asked to give their voluntary permission to fill out a questionnaire on possible erectile dysfunction.

The questionnaire consists of two parts: Part 1 is the IIEF (International Index of Erectile Function) questionnaire and Part 2 is an additional questionnaire. The included patients have to fill out these questionnaires two times; once at the beginning at a diabetic year program visit and a second time one year later at the next diabetic year program consultation.

The patients will also be asked to give their permission for using their results of the routine diabetic year program for scientific research.

ELIGIBILITY:
Inclusion Criteria:

* Male diabetic patients
* Age older than 18 years

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-05; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Documentation of the prevalence of erectile dysfunction in the diabetic convention
Increase the awareness of diabetologist for erectile dysfunction
Relation of erectile dysfunction with metabolic parameters
Relation of erectile dysfunction with sex steroids

SECONDARY OUTCOMES:
Adjustment of the systematic follow-up of diabetic complications.
Optimalisation of the healthcare for diabetic patients, so that the quality of life for male diabetic patients can be improved

CONTACTS AND LOCATIONS:
Overall Officials: Guy T'Sjoen, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be